CLINICAL TRIAL: NCT06733948
Title: Chemoradiotherapy With and Without Dental Stent for Taste Protection in Patients With Nasopharyngeal Carcinoma: a Randomized Controlled Trial
Brief Title: ChemoRT With and Without Dental Stent for Taste Protection in NPC Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NPC Dental Stent
Record Dates: First submitted 2024-09-16; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal cancer; dental stent; nasopharyngeal carcinoma; chemogustrometry; taste test; chemoradiation
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients are randomly assigned in a 1:1 ratio to Arm 1 and Arm 2. A web-based number generator will be used to generate random allocation lists using block sizes n =4 each. The treatment assignation is not masked. Subjects in the intervention group will receive the addition of dental stent to their radical concurrent chemoradiation, while those in the control group will receive radical concurrent chemoradiation with no dental stent. The process is not blinded to patient and investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Radiotherapy with dental stent +/- Concurrent systemic therapy
  Interventions: Device: Dental stent
- Control (Other): Radiotherapy with no dental stent +/- Concurrent systemic therapy
  Interventions: Other: No dental stent

INTERVENTIONS:
Device: Dental stent — Dental stent is personalised device for tongue depressing and immobilisation during RT. The aims are to reduce unnecessary RT doses to adjacent non-target healthy tissue, including the tongue, adjacent oral mucosa, parotid glands/ submandibular glands, and temporomandibular joints. Dentists will take impression of the teeth on moulds, and measure the height to raise the bite, the stent is then fabricated as methyl methacrylate resin in the dental laboratory. The resin base extends to the tongue and a flat plate depresses the tongue. This device will be placed before each RT fraction.
  Arms: Arm 1
Other: No dental stent — No dental stent used during chemoradiation treatment
  Arms: Control

SUMMARY:
Primary objective:

Evaluate and compare incidence of acute and long-term taste dysfunction in chemoradiation plus dental stent group vs. chemoradiation group, using objective-measured taste strip test, and patient-reported taste ability and toxicity.

Secondary objectives:

1. Evaluate and compare incidence of acute and long-term toxicities (excluding taste) and patient-reported quality of life between chemoradiation plus dental stent group and chemoradiation group.
2. Evaluate and compare tumor response, overall survival, and failure-free survival between chemoradiation plus dental stent group and chemoradiation group.
3. Analyze dosimetric parameters of taste bud bearing tongue mucosa, ipsilateral/ contralateral parotid and submandibular glands extracted from RT plans and correlate with taste impair

DETAILED DESCRIPTION:
This study is a phase II randomized control trial assessing the efficacy of adding a dental stent for sparing the taste bud and protect the taste sensation in NPC patients undergoing chemoradiation. The enrolled participants will be randomized to add a personalized dental stent during the radical chemoradiation to nasopharynx and neck using IMRT technique. Chemoradiation must begin no later than 4 weeks from the time of recruitment, although treatment as early as possible is highly encouraged.

A total of 50 patients (25 patients each arm) will be accrued to assess the potential benefit and safety of the said dental stent to standard chemoradiation.

All participants will be followed up as follows:

1. One visit before induction chemotherapy (if any)
2. One visit within 6 weeks before RT
3. Weekly during treatment and at the end of treatment (6-7 visits depending on treatment schedule),
4. One visit at 4 weeks post treatment (with +/-2 weeks window period)
5. One visit at 12 weeks post treatment (with +/- 4 weeks window period)
6. One visit at 26 weeks post treatment (with +/-4 weeks window period) and
7. One visit at 52 weeks post treatment (with +/-4 weeks window period) to review their general condition, toxicities, and long-term treatment efficacy and safety profile.

The assessment of taste sensation using subjective questionnaires, alongside objective measures using taste strip tests are performed at baseline, the 12 weeks post treatment follow up and at the 52 weeks post treatment follow up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Patients newly diagnosed with histologically confirmed non-keratinizing NPC.
2. Patients with Tumours staged as T1-4N+/TxN0-3.
3. No sign of distant metastasis (M0).
4. Satisfactory performance status (i.e., Karnofsky Performance Status ≥ 70 or ECOG < 2)
5. Age 21 years or older.
6. Adequate bone marrow function by peripheral blood counts as demonstrated by the following laboratory values:

   1. ≥ 3 × 109/L leucocytes
   2. ≥ 1.5 × 109/L neutrophils
   3. ≥ 9 g/dL of haemoglobin, and
   4. ≥ 100 × 109/L platelets.
7. Normal liver function demonstrated by the following laboratory values:

   1. Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) concentrations of < 1.5x upper limit of normal (ULN)
   2. Alkaline phosphatase (ALP) concentration < 2.5x ULN
   3. Bilirubin < ULN.
8. Renal function: Creatinine clearance at ≥60 mL/min
9. Able to provide informed consent

7. Induction chemotherapy before radical chemoradiation to nasopharynx and neck is permissible if no disease progression after induction chemotherapy

Exclusion Criteria:

1. Edentulous patients
2. Extensive crown/ implant work to the teeth
3. Patients having basaloid squamous cell carcinoma or WHO keratinizing squamous cell carcinoma.
4. Patients who suffered from previous malignancies, except adequately treated basal cell or squamous cell skin cancer, and in-situ cervical cancer.
5. Received RT previously (except for non-melanomatous skin cancers outside the intended RT treatment area)
6. Patients who received previous surgery (except diagnostic) or chemotherapy for the primary tumours or lymph nodes or history of glossectomy.
7. Patient who had a prior diagnosis of diseases effecting saliva secretion or causing salivary glands impairment (i.e., Sjogren's syndrome, iodine cancer treatment), had a reported history of abnormal sense of taste or eating disorders.
8. Current heavy smokers (smoke > 1 pack/day) or previous heavy smokers (stopped smoking less than 2 years and had smoked > 1 pack/day).
9. Patients suffering from any severe intercurrent disease, which may incur unacceptable risk or negatively affect trial compliance. For example, unstable cardiac disease necessitating treatment, chronic hepatitis renal disease, poorly controlled diabetes (fasting plasma glucose greater 1.5x upper limit of normal), and emotional disturbance.
10. Pregnant or lactating women.
11. Inability to attend the full course of RT or planned follow-up/survey responses.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Patient-assessed taste impairment using the QLQ-HN43 module | From baseline to 52 weeks post-RT
  Patient-assessed taste impairment measured on 4-point verbal rating scale, ranging from none to severe using the QLQ-HN43 module.
Taste impairment assessed on NCI CTCAE version 5.0 grading | From baseline to 52 weeks post RT
  Taste alterations (dysgeusia) will be graded between Grades 0 to 2.
Taste impairment measured on the STTA scale | From baseline to 52 weeks post-RT
  The STTA scale modified from the Late Effects Normal Tissue/Subjective Objective Management Analytic is a scoring system for taste acuity ranging from Grades 0 to 4
Objective testing using test strips | From baseline to 52 weeks post-RT
  Taste strips are a validated approach to assess taste ability for the five primary taste modalities - sweet, sour, salty, bitter, and umami.

SECONDARY OUTCOMES:
Acute toxicities (other than taste) graded according to NCI CTCAE V5.0 | From baseline to 52 weeks post-RT
  Other toxicities experienced by the patients during treatment. For example, dermatitis, mucositis, dry mouth will be graded according to the CTCAE V5.0 scales.
Acute toxicities (other than taste) graded according to the STTA scale | From baseline to 52 weeks post-RT
  Other toxicities experienced by the patients during treatment will be graded according to the STTA scale.
Patient-reported QoLs between the 2 groups according to EORTC modules QLQ-C30 and QLQ-HN43 | From enrollment to 52 weeks after the end of treatment
  EORTC QLQ-C30 and specific module for head and neck EORTC QLQ-HN43 will be used.
OS, FFS, distant FFS, and locoregional FFS between the 2 groups measured in years and months | From enrollment to 52 weeks after the end of treatment
  FFS was defined as the interval between randomization and distant failure, locoregional failure, or death from any cause, whichever happened first. OS was defined as the interval from randomization to death from any cause. The distant FFS was defined as the interval from randomization to the first distant metastasis. The locoregional FFS was defined as the interval from randomization to the first local or regional recurrence.
Dosimetry doses measured in Gy | From the first radiation therapy to the end of the radiation therapy at 6-7 weeks
  The mean, minimum, and maximum doses measured in gray (Gy) to the taste bud bearing tongue mucosa, the ipsilateral- and contralateral parotid and submandibular glands are extracted from the RT plans.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Cheo, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - Singapore Institute of Food and Biotechnology Innovation, Singapore
  - National University Hospital, Singapore